CLINICAL TRIAL: NCT01467024
Title: Evaluation of the MP Diagnostics HTLV Blot 2.4
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: MP Biomedicals, LLC (Industry)
Collaborators: Vital Systems Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: MP-EIA-HTLV-001B
Record Dates: First submitted 2011-10-31; First posted 2011-11-08 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-11

CONDITIONS: HTLV-I Infections; HTLV-II Infections; Human T-lymphotropic Virus 1; Human T-lymphotropic Virus 2; HTLV I Associated T Cell Leukemia Lymphoma; HTLV I Associated Myelopathies
Keywords: HTLV; Confirmatory; Supplemental; Blot; HTLV-I; HTLV-II
MeSH Terms: conditions — HTLV-I Infections; HTLV-II Infections; Leukemia-Lymphoma, Adult T-Cell; Paraparesis, Tropical Spastic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- EIA Negative: Blood donor specimens that tested non-reactive by previously licensed HTLV screening assay.
  Interventions: Other: CDPHL Algorithm
- EIA Repeat Reactive: Blood donor specimens that tested repeat reactive by previously licensed HTLV screening assay, but are unconfirmed.
  Interventions: Other: CDPHL Algorithm
- Known Positive: Blood donor specimens that tested repeat reactive with a licensed HTLV screening assay and have been confirmed through additional, unlicensed supplemental testing.
  Interventions: Other: CDPHL Algorithm

INTERVENTIONS:
Other: CDPHL Algorithm — Supplemental testing algorithm performed by the CDPHL.

SUMMARY:
The purpose of this study is:

1. To assess the validity and reproducibility of the MP Diagnostics HTLV Blot 2.4.
2. To conduct a sensitivity analysis of the HTLV Blot 2.4 using a known positive population.

DETAILED DESCRIPTION:
This is a retrospective study designed to assess the validity and reproducibility of the MP Diagnostics IVD device, the HTLV Blot 2.4 (MP Blot), in various populations. The study will be conducted at three geographical distinct locations.

The validity of the MP Blot will be assessed by calculating the following:

1. Percent negative agreement with CDPHL Algorithm on 200 EIA negative specimens
2. Percent positive agreement with CDPHL Algorithm on 200 EIA repeat reactive specimens

The sensitivity of the MP Blot will be evaluated by testing 200 known positive specimens. The study will be performed using three product lots at three clinical sites.

The reproducibility of the MP Blot will be assessed by testing two replicates of a three member panel at three clinical testing sites with each of three lots of product over multiple days by three operators.

ELIGIBILITY:
Inclusion Criteria:

* EIA Negative Population

  1. Male or female
  2. Completion of a health history evaluation for routine donor screening
  3. Willing and able to provide informed consent
  4. Negative screening assay results for all ARC screening assays
* EIA Repeat Reactive Population

  1. Male or female
  2. Completion of a health history evaluation for routine donor screening
  3. Willing and able to provide informed consent
  4. Previous RR result by bioMerieux ELISA, Abbott EIA, and / or Abbott ChLIA PRISM
* Known Positive Population

  1. Male or female
  2. Willing and able to provide informed consent
  3. Previous reactive screening test using either the bioMerieux ELISA, the Abbott EIA or the Abbott ChLIA PRISM, followed by supplemental testing

Exclusion Criteria:

* EIA Negative Population

  1. Inadequate sample volume for testing
  2. Unable to provide samples that meet the sample suitability requirements for testing
  3. Positive screening result for any infectious disease tested by ARC
* EIA Repeat Reactive Population

  1. Inadequate sample volume for testing
  2. Unable to provide samples that meet the sample suitability requirements for testing
  3. Positive result for HIV, HBV, HCV, or any other infectious disease
* Known Positive Population

  1. Unwilling or unable to provide informed consent
  2. Unable to provide adequate sample volume for testing
  3. Unable to provide samples that meet the sample suitability requirements for testing
  4. Positive result for HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All populations are from whole blood donors.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2011-11; Primary Completion 2012-01 (Estimated); Study Completion 2012-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Stramer, Ph.D, Principal Investigator — American National Red Cross
Locations (2):
- United States (2):
  - California Department of Public Health, Richmond, California
  - LABS, Inc, St Louis, Missouri